CLINICAL TRIAL: NCT06379893
Title: A Prospective Real-World Evidence Study Evaluating the Effects of Voltaren Use on Mobility and Quality of Life in Participants With Knee Osteoarthritis (OA) Pain
Brief Title: A Real-World Evidence Study to Evaluate the Effects of Voltaren Use on Mobility and Quality of Life in Participants With Knee Osteoarthritis Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300128; 2024-510839-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voltaren Gel (Experimental): Participants will use Voltaren Gel topically, applied daily as per label and leaflet instructions for up to 21 days. Participants will be instructed to wear Actigraph device on the wrist as per label, leaflet or site-specific instructions post training throughout the day for up to 21 days.
  Interventions: Drug: Voltaren Gel

INTERVENTIONS:
Drug: Voltaren Gel — Diclofenac sodium gel in 3 different concentrations as- Diclofenac sodium 1%, 1.16% and 2.32% whichever was available in the given region.

SUMMARY:
The purpose of this study is to investigate how topical diclofenac use can improve functional mobility and physical activity primarily, as well as other quality-of-life (QoL) parameters such as sleep, mood, and engagement in daily activities in participants with knee OA.

DETAILED DESCRIPTION:
This prospective open-label, single-arm, multi-country (United States [US] and European Union [EU]) real-world evidence study will be conducted in a hybrid form and will focus on assessing the impact of Voltaren Gel on functional mobility and QoL in individuals with mild/nonserious OA of the knee. Participants will be required to be physically present at the study site for screening, end of baseline and end of study visits. The remaining treatment will be conducted in a remote manner (for example, at home) to observe the real-world usage of Voltaren Gel. This study will utilize a research-grade validated wearable device: Actigraph, to accurately measure objective changes in functional mobility. Sufficient participants will be screened to enroll approximately 195 participants to ensure that around 147 of these participants will successfully complete the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is male or female who, at the time of screening, is between the ages of 40 and 85 years, inclusive.
* A participant who is willing and able to comply with scheduled visits, on-label Voltaren Gel use plan, and other study procedures.
* A participant willing to wear Actigraph continuously 24/7 for the study period.
* A participant in good general and mental health.
* A participant with diagnosed knee mild/non-serious osteoarthritis, proven via radiological evidence collected within the last 3 years.
* A participant with self-reported knee pain, with a score of greater than or equal to (>=) 40 millimeters (mm) less than or equal to (<=)70mm on the pain intensity visual analogue scale at the time of Informed Consent Form (ICF) signature.
* A participant willing to use Voltaren Gel for up to 3 weeks.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 1 month prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant with confirmed rheumatologic disease
* A participant who has experienced trauma to the knee within the last 2 months that resulted in pain and/or swelling.
* A participant that has been administered local steroids or other Non-steroidal anti-inflammatory drugs (NSAIDs) injections to the knee within the last 3 months.
* A participant with recent history of major knee injury or surgery.
* A participant with knee skin area pathological condition which prevents application of product to the skins. Conditions such as: open skin wounds, infections, inflammations, or exfoliative dermatitis conditions.
* A participant with conditions not limited to the following: Gastrointestinal diseases, asthma, hypertension, myocardial infarction, thrombotic events, stroke, congestive heart failure, impaired renal function, or liver disease as judged by investigator or Site Staff.
* A participant diagnosed with other relevant medical conditions (example, psychiatric, neurological).
* A participant who takes medication relating to above conditions, such as tricyclic antidepressants or anticonvulsants.
* A participant with an active infection.
* A participant who is pregnant, lactating, or plan to be pregnant or lactating during the study.
* A participant with use of aspirin, Oral NSAIDs, topical treatment with any NSAIDs, warfarin, Angiotensin-converting enzyme (ACE) inhibitors, cyclosporine, diuretics, lithium or methotrexate, corticosteroids, or other anticoagulant therapy within 30 days of study.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients, including hypersensitivity to NSAIDs and aspirin triad.
* A participant with any other acute or chronic illness that could compromise the integrity of study data or place the participant at risk by participating in the study.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (2):
  - Tandem Clinical Research, Marrero, Louisiana
  - Quality Research Inc, San Antonio, Texas
- Poland (6):
  - Vitamed Gałaj I Cichomski sp.j., Bydgoszcz
  - Centrum Medyczne Lukamed., Chojnice
  - Silmedic sp. z o.o., Katowice
  - Santa Sp. z o.o. Santa Familia PTG Lodz, Lodz
  - Centrum Badawcze Panaceum Agnieszka Brzezicka, Magdalena Lenkiewicz Sp z .o.o, Malbork
  - Specjalistyczny Osrodek Lecziczo Badawczy (SOLB) Zbgniew Żęgota, Ostróda

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in the United States (US) and 6 centers in the European Union (EU) (Poland).
Pre-assignment Details: A total of 214 participants were screened during study of which 196 participants were enrolled and received Voltaren Gel. A total of 194 participants completed the study.
Groups:
- Voltaren Gel: Participants used Voltaren Gel containing diclofenac sodium, topically, applied daily as per label and leaflet instructions for up to 21 days. Participants were instructed to wear Actigraph device on the wrist as per label, leaflet or site-specific instructions post training throughout the day for up to 21 days.
Period: Overall Study
Arm/Group | Voltaren Gel
Started | 196
Completed | 194
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Sponsors' decision | 1

BASELINE CHARACTERISTICS:
Population: The enrolled population included all participants who met the inclusion/exclusion criteria as recorded on the 'Participant Eligibility: Inclusion/Exclusion Criteria' electronic case report form (eCRF) page.
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 188
  More than one race | 1
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Only participants in the US were required to provide ethnicity and missing data refers to participants outside of the US.
  Participants
    Hispanic or Latino | 19
    Not Hispanic or Latino | 20
    Missing | 157

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Minutes of Moderate and Vigorous Physical Activity (MVPA) at Week 1
Description: The average minutes of MVPA were measured through a connected activity tracker (Actigraph device) worn by the participants to evaluate the effects of Voltaren Gel on physical activity. A mixed model with repeated measures (MMRM) was used to analyse the change from Baseline in MVPA average minutes. Change from Baseline was calculated by subtracting the Baseline average MVPA value from the average MVPA value at Week 1. Baseline value was calculated as the sum of minutes of MVPA over the Baseline period divided by duration of Baseline period, where Baseline period was the number of non-missing days between Day -6 and Day 0. A positive change from Baseline indicated improvement. Modified Intent-To-Treat (mITT) population included all participants who met the inclusion/exclusion criteria, who used study product at least once and had data from at least one post Baseline quality of life (QoL) questionnaire to support at least one of the secondary endpoint assessments.
Time Frame: Baseline and Week 1
Population: mITT Population. This study was designed as a single-arm real-world evidence (RWE) study to evaluate the effectiveness of Voltaren gel. There was no intention to compare the effectiveness of the three formulations within the population; therefore, all participants were analyzed as a single group. The reported results apply to the entire study population ("all groups") because there were no separate Arms/Groups in the study design.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
minutes
  Baseline | 249.2 (92.99)
  Change from Baseline at Week 1 | 14.2 (53.54)
Statistical Analysis 1: Comparison: Voltaren Gel; Change From Baseline at Week 1; Test type: Superiority; p < 0.001, MMRM; Least Square Means = 15.6, 95% CI 2-sided [8.3 to 22.8]

2. Primary Outcome: Change From Baseline in the Average Minutes of MVPA at Week 2
Description: The average minutes of MVPA were measured through a connected activity tracker (Actigraph device) worn by the participants to evaluate the effects of Voltaren Gel on physical activity. A MMRM was used to analyse the change from Baseline in MVPA average minutes. Change from Baseline was calculated by subtracting the Baseline average MVPA value from the average MVPA value at Week 2. Baseline value was calculated as sum of minutes of MVPA over the Baseline period divided by duration of Baseline period, where Baseline period was the number of non-missing days between Day -6 and Day 0. A positive change from Baseline indicated improvement.
Time Frame: Baseline and Week 2
Population: mITT population. This study was designed as a single-arm RWE study to evaluate the effectiveness of Voltaren gel. There was no intention to compare the effectiveness of the three formulations within the population; therefore, all participants were analyzed as a single group. The reported results apply to the entire study population ("all groups") because there were no separate Arms/Groups in the study design.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
minutes
  Baseline | 249.2 (92.99)
  Change from Baseline at Week 2 | 10.7 (60.93)
Statistical Analysis 1: Comparison: Voltaren Gel; Change From Baseline at Week 2; Test type: Superiority; p = 0.001, MMRM; Least Square Means = 13, 95% CI 2-sided [5.2 to 20.9]

3. Primary Outcome: Change From Baseline in the Average Minutes of MVPA at Week 3
Description: The average minutes of MVPA were measured through a connected activity tracker (Actigraph device) worn by the participants to evaluate the effects of Voltaren Gel on physical activity. A MMRM was used to analyse the change from Baseline in MVPA average minutes. Change from Baseline was calculated by subtracting the Baseline average MVPA value from the average MVPA value at Week 3. Baseline value was calculated as sum of minutes of MVPA over the Baseline period divided by duration of Baseline period, where Baseline period was the number of non-missing days between Day -6 and Day 0. A positive change from Baseline indicated improvement.
Time Frame: Baseline and Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
minutes
  Baseline | 249.2 (92.99)
  Change from Baseline at Week 3 | -0.8 (71.08)
Statistical Analysis 1: Comparison: Voltaren Gel; Change From Baseline at Week 3; Test type: Superiority; p = 0.653, MMRM; Least Square Means = 2.1, 95% CI 2-sided [-7.1 to 11.3]

4. Secondary Outcome: Change From Baseline in Daily Average Number of Steps Taken at Weeks 1, 2 and 3
Description: Daily average number of steps taken were measured through a connected activity tracker (Actigraph device) worn by the participants to evaluate the effects of Voltaren Gel on functional mobility. MMRM was used to analyse the change from Baseline in daily average number of steps taken. Change from Baseline was calculated by subtracting the average number of steps taken at Baseline from the average number of steps taken at each indicated post-Baseline timepoint. Baseline value was calculated as the sum of steps taken over the Baseline period divided by duration of Baseline period, where Baseline period was the number of non-missing days between Day -6 and Day 0. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
steps
  Baseline | 13826.5 (5076.05)
  Change from Baseline at Week 1 | 602.3 (2930.69)
  Change from Baseline at Week 2 | 323.1 (3515.66)
  Change from Baseline at Week 3 | -57.1 (3826.57)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p = 0.001, MMRM; Least Square Means = 707, 95% CI 2-sided [278.9 to 1135]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p = 0.040, MMRM; Least Square Means = 487.3, 95% CI 2-sided [22 to 952.6]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p = 0.603, MMRM; Least Square Means = 130.8, 95% CI 2-sided [-365.6 to 627.2]

5. Secondary Outcome: Change From Baseline in Ratio of Sedentary/Non-sedentary Time at Weeks 1, 2 and 3
Description: Sedentary/non-sedentary time was measured using a connected activity tracker (Actigraph device) worn by the participants to evaluate the effects of Voltaren Gel on functional mobility. Ratio of sedentary/non-sedentary time was calculated as = Total number of minutes defined as sedentary behaviour divided by Total number of non-sedentary behaviour minutes where number of non-sedentary behaviour minutes in the day was derived as the sum of light activity and MVPA. Change from Baseline was calculated by subtracting the Baseline ratio of sedentary/non-sedentary time from the ratio at each indicated post-Baseline timepoint. Baseline was defined as the number of non-missing days between Day -6 and Day 0. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: mITT population. Number analyzed is the number of participants with non-missing data at the indicated timepoint. This study was designed as a single-arm RWE study to evaluate the effectiveness of Voltaren gel. There was no intention to compare the effectiveness of the three formulations within the population; therefore, all participants were analyzed as a single group. The reported results apply to the entire study population ("all groups") as there were no separate Arms in the study design.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
ratio
  Baseline | 1.984 (1.1595)
  Change from Baseline at Week 1 | -0.028 (0.5376)
  Change from Baseline at Week 2: number analyzed (Participants) | 187
  Change from Baseline at Week 2 | 0.003 (0.5571)
  Change from Baseline at Week 3: number analyzed (Participants) | 185
  Change from Baseline at Week 3 | 0.089 (0.6121)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p = 0.473, MMRM; Least Square Means = -0.028, 95% CI 2-sided [-0.105 to 0.049]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p = 0.835, MMRM; Least Square Means = 0.009, 95% CI 2-sided [-0.074 to 0.091]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p = 0.014, MMRM; Least Square Means = 0.110, 95% CI 2-sided [0.023 to 0.198]

6. Secondary Outcome: Change From Baseline in Gait Assessed Through Speed and Step Irregularity Measured Via Cadence at Weeks 1, 2 and 3
Description: Gait was assessed through speed and step irregularity measured via cadence using a connected activity tracker (Actigraph device) worn by the participants. Change from Baseline was calculated as by subtracting the average cadence at Baseline from the cadence at each indicated post-Baseline timepoint. Baseline was defined as the number of non-missing days between Day -6 and Day 0. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: steps per minute
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
steps per minute
  Baseline | 109.207 (6.8045)
  Change from Baseline at Week 1 | -0.149 (6.3135)
  Change from Baseline at Week 2 | -1.126 (11.7981)
  Change from Baseline at Week 3 | -1.751 (14.7336)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p = 0.261, MMRM; Least Square Means = 0.261, 95% CI 2-sided [-0.196 to 0.717]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p = 0.263, MMRM; Least Square Means = 0.249, 95% CI 2-sided [-0.188 to 0.685]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p = 0.854, MMRM; Least Square Means = 0.053, 95% CI 2-sided [-0.512 to 0.617]

7. Secondary Outcome: Change From Baseline in Gait Assessed Through Speed and Step Irregularity Measured Via Gait Speed at Weeks 1, 2 and 3
Description: Gait was assessed through speed and step irregularity measured via gait speed using a connected activity tracker (Actigraph device) worn by the participants. Change from Baseline was calculated by subtracting the average gait speed at Baseline from the Average gait speed at each indicated post-Baseline timepoint. Baseline was defined as the number of non-missing days between Day -6 and Day 0. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: mITT population. Overall number analyzed is the number of participants with data available for analyses of this outcome measure. This study was designed as a single-arm RWE study to evaluate the effectiveness of Voltaren gel. There was no intention to compare the effectiveness of the 3 formulations within the population; So, all participants were analyzed as a single group. The reported results apply to the entire study population (all groups) as there were no separate Arms in the study design.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 177
meters per second
  Baseline | 1.010 (0.1385)
  Change from Baseline at Week 1 | -0.007 (0.0809)
  Change from Baseline at Week 2 | -0.016 (0.1069)
  Change from Baseline at Week 3 | -0.016 (0.1401)

8. Secondary Outcome: Change From Baseline in Indices of Morning Stiffness Assessed Through Levels of Mobility 30 Minutes Post-wake at Weeks 1, 2 and 3
Description: Indices of morning stiffness were assessed through levels of mobility 30 minutes post-wake. Functional mobility was measured through a connected activity tracker (Actigraph device) worn by the participants. Daily morning stiffness 30 minutes post-wake was defined as the total vector magnitude counts from Actigraph device 30 minutes post-wake. Change from Baseline was calculated as = (Average morning stiffness 30 minutes post-wake at each indicated post-Baseline timepoint minus Average Baseline morning stiffness 30 minutes post-wake). Baseline was defined as the number of non-missing days between Day -6 and Day 0. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: mITT population. Overall number analyzed is the number of participants with data available for analyses of this outcome measure. Number analyzed is the number of participants with non-missing data at the indicated timepoint. This study was designed as a single-arm RWE study to evaluate the effectiveness of Voltaren gel. There was no intention to compare the effectiveness of the 3 formulations within the population. The reported results apply to the entire study population ("all groups").
Measure: Mean (Standard Deviation); unit: vector magnitude counts
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
vector magnitude counts
  Baseline | 75593.364 (44958.5420)
  Change from Baseline at Week 1: number analyzed (Participants) | 187
  Change from Baseline at Week 1 | 1969.758 (28283.0182)
  Change from Baseline at Week 2: number analyzed (Participants) | 186
  Change from Baseline at Week 2 | 2332.422 (28420.8109)
  Change from Baseline at Week 3: number analyzed (Participants) | 184
  Change from Baseline at Week 3 | -1893.342 (34458.1863)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p = 0.221, MMRM; Least Square Means = 2415.2, 95% CI 2-sided [-1466.3 to 6296.8]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p = 0.127, MMRM; Least Square Means = 3041.7, 95% CI 2-sided [-868.5 to 6951.9]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p = 0.314, MMRM; Least Square Means = -2428.7, 95% CI 2-sided [-7177.5 to 2320.1]

9. Secondary Outcome: Change From Baseline in Indices of Morning Stiffness Assessed Through Levels of Mobility 60 Minutes Post-wake at Weeks 1, 2 and 3
Description: Indices of morning stiffness were assessed through levels of mobility 60 minutes post-wake. Functional mobility was measured through a connected activity tracker (Actigraph device) worn by the participants. Daily morning stiffness 60 minutes post-wake was defined as the total vector magnitude counts from Actigraph device 60 minutes post-wake. Change from Baseline was calculated as = (Average morning stiffness 60 minutes post-wake at each indicated post-Baseline timepoint minus Average Baseline morning stiffness 30 minutes post-wake). Baseline was defined as the number of non-missing days between Day -6 and Day 0. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: mITT Population. Here, overall number analyzed is the number of participants with data available for analyses of this outcome measure. Number analyzed is the number of participants with non-missing data at the indicated timepoint. This study was designed as a single-arm RWE study to evaluate the effectiveness of Voltaren gel. There was no intention to compare the effectiveness of the 3 formulations within the population. The reported results apply to the entire study population ("all groups").
Measure: Mean (Standard Deviation); unit: vector magnitude counts
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
vector magnitude counts
  Baseline | 149034.401 (86661.4977)
  Change from Baseline at Week 1: number analyzed (Participants) | 187
  Change from Baseline at Week 1 | 2891.276 (45249.4973)
  Change from Baseline at Week 2: number analyzed (Participants) | 186
  Change from Baseline at Week 2 | 2438.403 (48859.7477)
  Change from Baseline at Week 3: number analyzed (Participants) | 184
  Change from Baseline at Week 3 | -6734.944 (54957.9211)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p = 0.289, MMRM; Least Square Means = 3409.9, 95% CI 2-sided [-2911.4 to 9731.2]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p = 0.303, MMRM; Least Square Means = 3552.3, 95% CI 2-sided [-3240.4 to 10345.1]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p = 0.046, MMRM; Least Square Means = -7820.7, 95% CI 2-sided [-15512.8 to -128.5]

10. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Physical Function Subscale Score at Week 1, 2 and 3
Description: Participants completed the WOMAC questionnaire daily using eDiary. The WOMAC questionnaire consisted of 24 questions categorised in 3 subscales - Pain, Stiffness, Physical function. The physical function subscale consisted of 17 questions related to level of difficulty in performing functions, on average, during the last 48 hours scored on a 5-point Likert scale with scores ranging from 0 to 4, where score 0=none, 1=slight, 2=moderate, 3=severe, 4=extreme. Total WOMAC physical function subscale score was normalized on a 0 to 100 scale calculated as = (sum of raw score items)*1.47. Higher scores indicated more difficulty in performing physical functions. Change from Baseline was calculated by subtracting the normalized WOMAC subscale score at Baseline from the normalized WOMAC subscale score at each indicated post-Baseline timepoint. Baseline was defined as Day 0. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 176
score on a scale
  Baseline | 48.702 (12.9284)
  Change from Baseline at Week 1: number analyzed (Participants) | 165
  Change from Baseline at Week 1 | -8.677 (12.6188)
  Change from Baseline at Week 2: number analyzed (Participants) | 159
  Change from Baseline at Week 2 | -11.926 (14.0764)
  Change from Baseline at Week 3: number analyzed (Participants) | 167
  Change from Baseline at Week 3 | -15.644 (16.9641)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -8.392, 95% CI 2-sided [-10.196 to -6.588]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -11.882, 95% CI 2-sided [-13.946 to -9.818]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -15.929, 95% CI 2-sided [-18.320 to -13.537]

11. Secondary Outcome: MVPA on Each Day of the Study
Description: The average minutes of MVPA on each day were measured through a connected activity tracker (Actigraph device) worn by the participants to assess the functional mobility. Baseline was calculated as the average of MVPA values collected during the Baseline period, where Baseline period was the number of non-missing days between Day -6 and Day 0.
Time Frame: Baseline up to Day 21
Population: mITT population. Number analyzed is the number of participants with non-missing data at the indicated timepoint. This study was designed as a single-arm RWE study to evaluate the effectiveness of Voltaren gel. There was no intention to compare the effectiveness of the 3 formulations within the population; So, all participants were analyzed as a single group. The reported results apply to the entire study population (all groups) as there were no separate Arms in the study design.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 188
minutes
  Baseline | 249.2 (92.99)
  Day 1 | 274.1 (119.79)
  Day 2 | 268.4 (124.96)
  Day 3 | 259.3 (124.79)
  Day 4 | 270.8 (126.09)
  Day 5 | 255.8 (115.05)
  Day 6 | 255.1 (119.03)
  Day 7 | 260.4 (112.45)
  Day 8 | 264.2 (122.21)
  Day 9 | 258.0 (126.33)
  Day 10 | 266.5 (128.05)
  Day 11 | 262.9 (124.18)
  Day 12 | 252.0 (122.99)
  Day 13 | 261.3 (122.89)
  Day 14 | 254.3 (114.00)
  Day 15 | 254.6 (124.49)
  Day 16: number analyzed (Participants) | 187
  Day 16 | 250.3 (114.15)
  Day 17: number analyzed (Participants) | 187
  Day 17 | 251.1 (122.16)
  Day 18: number analyzed (Participants) | 187
  Day 18 | 253.8 (124.67)
  Day 19: number analyzed (Participants) | 187
  Day 19 | 239.1 (118.63)
  Day 20: number analyzed (Participants) | 187
  Day 20 | 244.0 (120.81)
  Day 21: number analyzed (Participants) | 185
  Day 21 | 107.8 (85.88)

12. Secondary Outcome: WOMAC Physical Function Subscale Score at Weeks 1, 2 and 3
Description: Physical function subscale score of the WOMAC questionnaire was used to study participant's perceived ability to exercise more regularly. It consisted of 17 questions related to the level of difficulty in performing functions, on average, during the last 48 hours scored on a 5-point Likert scale with scores ranging from 0 to 4, daily using eDiary where score 0=none, 1=slight, 2=moderate, 3=severe, 4=extreme. Total WOMAC physical function subscale score was normalized on a 0 to 100 scale calculated as = (sum of raw score items)*1.47. Higher scores indicated more difficulty in performing physical functions.
Time Frame: Week 1, Week 2 and Week 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 176
score on a scale
  Week 1: number analyzed (Participants) | 174
  Week 1 | 40.375 (14.7527)
  Week 2: number analyzed (Participants) | 169
  Week 2 | 37.072 (15.9130)
  Week 3 | 32.781 (17.2916)

13. Secondary Outcome: Change From Baseline in Self-reported Pain Intensity Assessed Through Numeric Rating Scale (NRS) at Weeks 1, 2 and 3
Description: Participants rated the pain intensity experienced by them daily within the eDiary, using NRS. NRS is an 11-point scale with scores ranging from 0 to 10 where score 0 = no pain, 1 = slight pain, 2-3 = mild pain, 4-6 = moderate pain, 7 = severe pain, 8 to 9 = extreme pain, 10=pain as bad as it could be. Higher scores indicated greater pain intensity. Change from Baseline was calculated by subtracting the Baseline NRS score from the NRS score at each indicated post-Baseline timepoint. Baseline was defined as Day 0. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 176
score on a scale
  Baseline | 5.7 (1.31)
  Change from Baseline at Week 1: number analyzed (Participants) | 166
  Change from Baseline at Week 1 | -1.5 (1.54)
  Change from Baseline at Week 2: number analyzed (Participants) | 162
  Change from Baseline at Week 2 | -1.9 (1.69)
  Change from Baseline at Week 3: number analyzed (Participants) | 169
  Change from Baseline at Week 3 | -2.6 (1.96)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -1.4, 95% CI 2-sided [-1.7 to -1.2]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -2, 95% CI 2-sided [-2.2 to -1.7]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -2.6, 95% CI 2-sided [-2.9 to -2.3]

14. Secondary Outcome: Change From Baseline in the WOMAC Total Score at Weeks 1, 2 and 3
Description: Participants completed the WOMAC questionnaire daily. The WOMAC questionnaire consisted of 24 questions each scored on a 5-point scale: 0=none, 1=slight, 2=moderate, 3=severe, 4=extreme. The WOMAC questionnaire was categorized in 3 subscales - Pain (5 questions, score ranges 0-20), Stiffness (2 questions, score ranges 0-8), Physical function (17 questions, score ranges 0-68). Each subscale score was normalized on a 0 to 100 scale calculated as: Pain subscale score= (sum of raw score items in dimension)*5; Stiffness subscale score= (sum of raw score items in dimension)*12.5; Physical function subscale score= (sum of raw score items in dimension)*1.47. WOMAC Total score = sum of the 3 normalized WOMAC subscale scores. Thus, WOMAC total score ranges from 0 to 300 with 0 being the best and 300 being the worst. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated post-Baseline timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 176
score on a scale
  Baseline | 147.040 (38.1349)
  Change from Baseline at Week 1: number analyzed (Participants) | 165
  Change from Baseline at Week 1 | -27.359 (38.7623)
  Change from Baseline at Week 2: number analyzed (Participants) | 159
  Change from Baseline at Week 2 | -36.062 (42.4964)
  Change from Baseline at Week 3: number analyzed (Participants) | 167
  Change from Baseline at Week 3 | -47.852 (49.4526)
Statistical Analysis 1: Comparison: Voltaren Gel; Change From Baseline at Week 1; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -26.529, 95% CI 2-sided [-31.929 to -21.129]
Statistical Analysis 2: Comparison: Voltaren Gel; Change From Baseline at Week 2; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -36.179, 95% CI 2-sided [-42.090 to -30.269]
Statistical Analysis 3: Comparison: Voltaren Gel; Change From Baseline at Week 3; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -48.834, 95% CI 2-sided [-55.692 to -41.976]

15. Secondary Outcome: Change From Baseline in the WOMAC Pain Subscale Score at Weeks 1, 2 and 3
Description: The pain subscale of the WOMAC questionnaire consisted of 5 questions related to severity of pain experienced by the participant when walking, stair climbing, at night, at rest, weightbearing, on average, during the last 48 hours. Participants scored the questions on a 5-point Likert scale ranging from 0 to 4 daily using eDiary where score 0=none, 1=slight, 2=moderate, 3=severe, 4=extreme. The total pain subscale score was normalized on a 0 to 100 scale calculated as = (sum of raw score items in dimension)*5. Higher scores indicated more pain. Change from Baseline was calculated by subtracting the Baseline normalized WOMAC pain subscale score from the normalized score at each indicated post-Baseline timepoint. Baseline was defined as Day 0. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 176
score on a scale
  Baseline | 48.196 (13.2952)
  Change from Baseline at Week 1: number analyzed (Participants) | 166
  Change from Baseline at Week 1 | -9.458 (13.7044)
  Change from Baseline at Week 2: number analyzed (Participants) | 160
  Change from Baseline at Week 2 | -12.422 (14.5893)
  Change from Baseline at Week 3: number analyzed (Participants) | 169
  Change from Baseline at Week 3 | -16.383 (16.6274)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -9.213, 95% CI 2-sided [-11.011 to -7.415]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -12.570, 95% CI 2-sided [-14.519 to -10.621]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -16.408, 95% CI 2-sided [-18.669 to -14.146]

16. Secondary Outcome: Change From Baseline in the WOMAC Stiffness Subscale Score at Weeks 1, 2 and 3
Description: The stiffness subscale of the WOMAC questionnaire consisted of 2 questions related to severity of stiffness experienced by the participant at morning and during the day, on average, during the last 48 hours. Participants scored the questions on a 5-point Likert scale with scores ranging from 0 to 4 daily using eDiary, where score 0=none, 1=slight, 2=moderate, 3=severe, 4=extreme. The total stiffness subscale score for was normalized on a 0 to 100 scale calculated as = (sum of raw score items in dimension)*12.5. Higher scores indicated more stiffness. Change from Baseline was calculated by subtracting the Baseline normalized WOMAC stiffness subscale score from the normalized score at each indicated post-Baseline timepoint. Baseline was defined as Day 0. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 1, Week 2 and Week 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 176
score on a scale
  Baseline | 50.142 (16.7965)
  Change from Baseline at Week 1: number analyzed (Participants) | 165
  Change from Baseline at Week 1 | -9.242 (18.6173)
  Change from Baseline at Week 2: number analyzed (Participants) | 160
  Change from Baseline at Week 2 | -11.719 (19.2063)
  Change from Baseline at Week 3: number analyzed (Participants) | 169
  Change from Baseline at Week 3 | -15.680 (20.6853)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Week 1; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -8.912, 95% CI 2-sided [-11.401 to -6.423]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Week 2; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -11.699, 95% CI 2-sided [-14.177 to -9.221]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Week 3; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -16.166, 95% CI 2-sided [-18.858 to -13.473]

17. Secondary Outcome: Change From Baseline in Sleep/Alertness Assessed Using Karolinska Sleepiness Scale (KSS) at Days 7, 14 and 21
Description: KSS measured the subjective level of sleepiness/alertness during the day. Participants rated how sleepy or alert they were feeling using KSS with scores ranging from 1 to 9 where 1 = extremely alert, 2 = very alert, 3 = alert, 4 = fairly alert, 5 = neither alert nor sleepy, 6 = some signs of sleepiness, 7 = sleepy, but no efforts to keep alert, 8 = sleepy, some efforts to keep alert, 9 = very sleepy, great effort to keep alert, fighting sleep. Higher scores indicated greater sleepiness. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated post-Baseline timepoint. Baseline was defined as Day 0. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Day 7, Day 14, and Day 21
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 176
score on a scale
  Baseline | 3.9 (1.60)
  Change from Baseline at Day 7: number analyzed (Participants) | 166
  Change from Baseline at Day 7 | -0.2 (1.56)
  Change from Baseline at Day 14: number analyzed (Participants) | 163
  Change from Baseline at Day 14 | -0.2 (1.70)
  Change from Baseline at Day 21: number analyzed (Participants) | 169
  Change from Baseline at Day 21 | -0.4 (1.66)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Day 7; Test type: Superiority; p = 0.237, MMRM; Least Square Means = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Day 14; Test type: Superiority; p = 0.071, MMRM; Least Square Means = -0.2, 95% CI 2-sided [-0.4 to 0.0]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Day 21; Test type: Superiority; p < 0.001, MMRM; Least Square Means = -0.4, 95% CI 2-sided [-0.6 to -0.2]

18. Secondary Outcome: Change From Baseline in Health-related QoL Assessed Using EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Questionnaire at Days 7, 14, and 21
Description: Health-related QoL of participants was assessed using the EQ-5D-5L questionnaire. It consisted of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with 5 response levels for each dimension where Level 1 = no problems, Level 2 = slight problems, Level 3 = moderate problems, Level 4 = severe problems, Level 5 = unable to perform activities/extreme problems. Participants were asked to indicate their health by ticking the box next to the most appropriate response level for each dimension. The response levels were used to derive a health index score based on the Crosswalk Value Set for the United States ranging from less than 0 (worst imaginable health) to 1 (best imaginable health) where higher scores indicated better health. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. Baseline was defined as Day 0. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Days 7, 14 and 21
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voltaren Gel
Number analyzed (Participants) | 174
score on a scale
  Baseline | 0.67 (0.124)
  Change from Baseline at Day 7: number analyzed (Participants) | 155
  Change from Baseline at Day 7 | 0.04 (0.098)
  Change from Baseline at Day 14: number analyzed (Participants) | 154
  Change from Baseline at Day 14 | 0.05 (0.097)
  Change from Baseline at Day 21: number analyzed (Participants) | 164
  Change from Baseline at Day 21 | 0.07 (0.111)
Statistical Analysis 1: Comparison: Voltaren Gel; Change from Baseline at Day 7; Test type: Superiority; p < 0.001, MMRM; Least Square Means = 0.04, 95% CI 2-sided [0.02 to 0.05]
Statistical Analysis 2: Comparison: Voltaren Gel; Change from Baseline at Day 14; Test type: Superiority; p < 0.001, MMRM; Least Square Means = 0.05, 95% CI 2-sided [0.04 to 0.07]
Statistical Analysis 3: Comparison: Voltaren Gel; Change from Baseline at Day 21; Test type: Superiority; p < 0.001, MMRM; Least Square Means = 0.07, 95% CI 2-sided [0.05 to 0.09]

ADVERSE EVENTS:
Time Frame: From signing of informed consent form up to end of study (up to approximately 28 days)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A serious AE (SAE) was a particular category of an AE where the adverse outcome was serious.
Arm/Group | Voltaren Gel
All-Cause Mortality (participants affected / at risk) | 0/196
Serious Adverse Events (participants affected / at risk) | 0/196
Other Adverse Events (participants affected / at risk) | 17/196
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voltaren Gel (N=196)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Ear infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT06379893/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT06379893/SAP_001.pdf